CLINICAL TRIAL: NCT00763906
Title: Continuous Administration of Norepinephrine Assisted by Fuzzy Logic Assisted Control in Septic Shock Patients
Brief Title: Norepinephrine Weaning in Septic Patients
Acronym: CATECHOFLOU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DH/JF-11-2002
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Septic Shock
Keywords: septic shock; fuzzy logic; norepinephrine weaning
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Patients were assigned to norepinephrine infused at the clinician's discretion.
  Interventions: Device: norepinephrine infused at the clinician's discretion
- 2 (Active Comparator): Patients were assigned to norepinephrine infused under computerized fuzzy logic control.
  Interventions: Device: norepinephrine infused under computerized fuzzy logic control

INTERVENTIONS:
Device: norepinephrine infused at the clinician's discretion
  Arms: 1
Device: norepinephrine infused under computerized fuzzy logic control
  Arms: 2

SUMMARY:
The weaning rate of vasopressors drugs is usually chosen empirically by the clinician in critically patients. The investigators applied fuzzy logic principles to modify intravenous norepinephrine infusion rates during norepinephrine infusion in septic patients in order to reduce the duration of shock. The investigators goal was to reduce the duration of poorly controlled hemodynamic status.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock

Exclusion Criteria:

* Less than 18 years
* Pregnancy
* Weight above 135 kg
* Requirement for continuous epinephrine infusion
* Severe head injury, stroke, a comatose state following cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Primary Completion 2006-11 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Time to shock resolution defined as cessation of vasopressor support

SECONDARY OUTCOMES:
28 days survival, total amount of norepinephrine infused, duration of mechanical ventilation, and length of stay in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Réanimation, Bobigny, Seine-Saint-Denis, France

REFERENCES:
- [Derived] Merouani M, Guignard B, Vincent F, Borron SW, Karoubi P, Fosse JP, Cohen Y, Clec'h C, Vicaut E, Marbeuf-Gueye C, Lapostolle F, Adnet F. Norepinephrine weaning in septic shock patients by closed loop control based on fuzzy logic. Crit Care. 2008;12(6):R155. doi: 10.1186/cc7149. Epub 2008 Dec 9. PMID 19068113